CLINICAL TRIAL: NCT04568915
Title: Comparison Between Dry Needling and Maitland Joint Mobilization Techniques in Patients With Myofacial Chronic Neck Pain
Brief Title: Dry Needling and Maitland Joint Mobilization Techniques in Patients With Myofacial Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS-OMPT/Spring19/030 Momna; Momna Ghaffar (Other: Riphah)
Record Dates: First submitted 2020-09-25; First posted 2020-09-29 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Myofacial Pain; Neck Pain
Keywords: Neck Pain; Myofacial Pain
MeSH Terms: conditions — Facial Pain; Neck Pain | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry Needling-Group (Experimental): Tens, Stretching, Strengthening(girdle), Neck Isometrics, DN
  Interventions: Other: Dry Needling
- Maitland-Group (Active Comparator): Tens Stretching, Strengthening(girdle), Neck Isometrics, Maitland joint mobilization
  Interventions: Other: Maitland Mobilization

INTERVENTIONS:
Other: Dry Needling — TENS 10 minutes, Stretching, Strengthening(girdle),Neck Isometrics, DN
  Arms: Dry Needling-Group
Other: Maitland Mobilization — TENS 10 minutes, Stretching, Strengthening(girdle),Neck Isometrics, Maitland joint mobilization
  Arms: Maitland-Group

SUMMARY:
The purpose of my research is to compare the effects of dry needling and Maitland mobilization in chronic myofacial neck pain

DETAILED DESCRIPTION:
To distinguish which technique is most effective in pain reduction and range gain because in chronic cases there is involvement of fascia, muscles and joints due to prolonged stress on any of the component affecting the other. Hence, the study will help to design a treatment plan with more accurate intervention. After sample collection according to selection criteria treatment sessions will be given to both groups for 6 weeks. Data will be collected at baseline, then after 2 weeks, 4 weeks and at 8th week. Tools for data collection are Visual analogue scale, Neck Disability Index and Goniometer. For statistical analysis SPSS 22 will be used. Intra group difference will be calculated by repeated measurement ANOVA / Friedman test and inter group analysis will be done by Independent sample t test. Descriptive data will be expressed in terms of frequency and proportions.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral pain involving the upper trapezius and elevator muscle of the scapula;
* Duration of pain of at least 3 months;
* A pain intensity corresponding to at least 20 mm on a 100 mm visual analogue scale (VAS)
* Neck pain with symptoms provoked by either neck postures or neck movement;
* Pain localized at least in the cervical and occipital regions but not in the orofacial region;
* Neck disability index (NDI) greater than or equal to 15 points;
* Restricted cervical range of movements (flexion, extension, rotation, and sidebending); (i) Presence of bilateral MTrPs in upper trapezius and levator scapulae muscles

Exclusion Criteria:

* Any signs, symptoms, or history of the following diseases:
* Orofacial pain and temporo-mandibular disorders
* A history of traumatic injuries (e.g., contusion, fracture, and whiplash injury);
* Systemic diseases such as fibromyalgia, systemic erythematous lupus, and arthritis; (d) Neurologic disorders (e.g., trigeminal neuralgia or occipital neuralgia);
* Concomitant medical diagnosis of any primary headache (tension type or migraine);
* Unilateral neck pain;
* Cervical spine surgery;
* Clinical diagnosis of cervical radiculopathy or myelopathy;
* Needle phobia;
* History of previous physical therapy intervention for the cervical region in last 6 months.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2020-06-28 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale NPRS | 4 months
  The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).
Range of Motion | 4 months
  Standard Goniometer will be used.Higher score shows improvement.
Disability | 4 months
  Scoring: For each section the total possible score is 5: if the first statement is marked the section score = 0, if the last statement is marked it = 5. If all ten sections are completed the score is calculated as follows: Example:16 (total scored) 50 (total possible score) x 100 = 32% If one section is missed or not applicable the score is calculated: 16 (total scored) 45 (total possible score) x 100 = 35.5% Minimum Detectable Change (90% confidence): 5 points or 10 %points

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Shabbir, PHD, Principal Investigator — Riphah International University
Locations (1):
- Riphah IU, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gross A, Miller J, D'Sylva J, Burnie SJ, Goldsmith CH, Graham N, Haines T, Bronfort G, Hoving JL. Manipulation or mobilisation for neck pain. Cochrane Database Syst Rev. 2010 Jan 20;(1):CD004249. doi: 10.1002/14651858.CD004249.pub3. PMID 20091561
- [Background] Davidoff RA. Trigger points and myofascial pain: toward understanding how they affect headaches. Cephalalgia. 1998 Sep;18(7):436-48. doi: 10.1046/j.1468-2982.1998.1807436.x. PMID 9793695
- [Background] Borg-Stein J, Simons DG. Focused review: myofascial pain. Arch Phys Med Rehabil. 2002 Mar;83(3 Suppl 1):S40-7, S48-9. doi: 10.1053/apmr.2002.32155. PMID 11973695
- [Background] Campa-Moran I, Rey-Gudin E, Fernandez-Carnero J, Paris-Alemany A, Gil-Martinez A, Lerma Lara S, Prieto-Baquero A, Alonso-Perez JL, La Touche R. Comparison of Dry Needling versus Orthopedic Manual Therapy in Patients with Myofascial Chronic Neck Pain: A Single-Blind, Randomized Pilot Study. Pain Res Treat. 2015;2015:327307. doi: 10.1155/2015/327307. Epub 2015 Nov 10. PMID 26640708
- [Background] Blanpied PR, Gross AR, Elliott JM, Devaney LL, Clewley D, Walton DM, Sparks C, Robertson EK. Neck Pain: Revision 2017. J Orthop Sports Phys Ther. 2017 Jul;47(7):A1-A83. doi: 10.2519/jospt.2017.0302. PMID 28666405
- [Background] Dunning J, Butts R, Mourad F, Young I, Flannagan S, Perreault T. Dry needling: a literature review with implications for clinical practice guidelines. Phys Ther Rev. 2014 Aug;19(4):252-265. doi: 10.1179/108331913X13844245102034. PMID 25143704
- [Background] Graff-Radford SB, Reeves JL, Jaeger B. Management of chronic head and neck pain: effectiveness of altering factors perpetuating myofascial pain. Headache. 1987 Apr;27(4):186-90. doi: 10.1111/j.1526-4610.1987.hed2704186.x. No abstract available. PMID 3597072
- [Background] Tekin L, Akarsu S, Durmus O, Cakar E, Dincer U, Kiralp MZ. The effect of dry needling in the treatment of myofascial pain syndrome: a randomized double-blinded placebo-controlled trial. Clin Rheumatol. 2013 Mar;32(3):309-15. doi: 10.1007/s10067-012-2112-3. Epub 2012 Nov 9. PMID 23138883